CLINICAL TRIAL: NCT02243514
Title: Intravascular Ultrasound Evaluation of the Renal Nerves Remodeling in Different Diseases
Brief Title: Intravascular Ultrasound Evaluation of Renal Nerves in Different Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Jing Huang, Professor and Vice Director, Department of Cardiology, The Second Affiliated Hospital of Chongqing Medical University
Other Study IDs: US-RNRE; NSFC81370440 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2014-09-16; First posted 2014-09-18 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Hypertension; Heart Failure
Keywords: Hypertension; Heart failure; Sympathetic hyperactivity; Renal nerve; Remodeling; Nerve remodeling
MeSH Terms: conditions — Hypertension; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood, urine, stool
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Resistant hypertension
- Essential hypertension
- Chronic heart failure
- Control

SUMMARY:
Sympathetic hyperactivity is a causal or a promoting factor in many diseases, under these conditions, some morphology changes due to the hyperactivity occur. Renal nerve is an important part in the autonomic nervous system regulation, especially in cardiovascular system, the modulation of the renal nerves used as a therapeutic strategy has been researched across the world. The purpose of this study is to evaluate and quantify the morphology changes in different diseases, make the modulation therapy more selective and effective.

DETAILED DESCRIPTION:
People eligible for this study will be divided into 4 groups according to the eligibility criteria(Resistant Hypertension Group,Essential Hypertension Group, Chronic Heart Failure Group and Control Group), about 15 objects for each, totally 60 objects are going to be recruited.

Before the intravascular ultrasound examination, ambulatory blood pressure, ECG, plasma catecholamine hormones, renin-angiotension-aldosterone, ect. will be measured. An intravascular ultrasound examination will be taken after all of these have been done.

ELIGIBILITY:
Inclusion Criteria:

1. Resistant hypertension group

   * blood pressure remains above goal in spite of the concurrent use of three or more anti-hypertensive agents(including a diuretic) at adequate doses.
   * agrees to have the study procedure(s) performed and additional procedures and evaluations
2. Essential hypertension group

   * systolic blood pressure ≥ 140 mmHg, diastolic blood pressure ≥ 90 mmHg, or current use of anti-hypertensive medication with a normal blood pressure or mean ambulatory blood pressure during the 24-hour≥130/80 mmHg.
   * not resistant to pharmacotherapy.
   * agrees to have the study procedure(s) performed and additional procedures and evaluations
3. Chronic heart failure group

   * New York Heart Association class II-III symptoms, or American College of Cardiology(ACC) / American Heart Association(AHA) heart failure classification B-C class of chronic heart failure.
   * currently or prior have the signs of heart failure, such as elevated jugular venous pressure, peripheral edema, pulmonary crepitations, ect.
   * Systolic left ventricular dysfunction as assessed by echocardiogram with left ventricular ejection fraction < 40%.
   * agrees to have the study procedure(s) performed and additional procedures and evaluations
4. Control group

   * no history of arterial hypertension, heart failure and diabetes
   * going to take a vascular interventional examination during hospitalization
   * agrees to have the study procedure(s) performed and additional procedures and evaluations

All patients have full capacity for civil conduct and agree to sign the Medical Informed Consent.

Exclusion Criteria:

* hemodynamically or anatomically significant renal artery stenosis.
* renal artery variation.
* renal artery diameter < 4 mm, trunk length < 20 mm.
* secondary hypertension with known causes and pseudo-hypertension.
* has experienced myocardial infarction, unstable angina pectoris, or cerebrovascular accident within 6 months.
* has an implantable cardioverter defibrillator (ICD) or pacemaker.
* requires respiratory support.
* is pregnant or planning to be pregnant.
* cardiovascular diseases with sever hemodynamic disorder.
* type 1 diabetes mellitus.
* currently enrolled in another investigational drug or device trial.
* civil disability or limited capacity for civil conduct.
* other conditions researchers considered unsuitable for enrolled in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients who are going to take a vascular interventional examination.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-02 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Number increase of Renal nerves in patients with sympathetic over-activity diseases | A duration of the whole research stage, an expected average of 1/2 year
  Total number of the renal nerve of each patient(automatic identification by the embedded software in the ultrasound imaging host/counting manually): Number of Nerve Bundles;
Area increase of Renal nerves in patients with sympathetic over-activity diseases | A duration of the whole research stage, an expected average of 1/2 year
  Total area of the renal nerve (measured by ultrasound imaging host) of each patient: square millimeter (mm²)=∑= Nerve 1(length*width)+ Nerve 2(length*width)+ ......+ Nerve n(length*width);
The increase of the ratio of nerve area/artery wall area in patients with sympathetic over-activity diseases. | A duration of the whole research stage, an expected average of 1/2 year
  1. Renal artery area of each patient (measured by ultrasound imaging host): Square millimeter (mm²);
  2. Renal arterial wall area (measured by ultrasound imaging host) of each patient: Square millimeter (mm²);
  3. Total area of the renal nerve/Total renal artery area: percentage (%);
  4. Total area of the renal nerve/Total renal arterial wall area: percentage (%);

SECONDARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events Related to The Intervention Procedure | Participants will be followed for the duration of the operation time, an expected average of 0.5-1 hours
  Renal arteriography will be carried out post operation to evaluate the possibility of renal artery injuries caused by this procedure, which including:
  1. Emerging renal artery dissection;
  2. Emerging renal artery stenosis, which will not improve by the intravascular injection of nitroglycerin;
  3. Emerging renal artery rupture or perforate;
  4. Contrast-induced nephropathy
  5. Any other complications related to this intervention procedure, such as catheter breakage, infection, hematoma ect.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Huang, MD, Principal Investigator — Dept. of Cardiology, the 2nd affiliated hospital of Chongqing Medical University
Locations (1):
- The 2nd Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Bhatt DL, Kandzari DE, O'Neill WW, D'Agostino R, Flack JM, Katzen BT, Leon MB, Liu M, Mauri L, Negoita M, Cohen SA, Oparil S, Rocha-Singh K, Townsend RR, Bakris GL; SYMPLICITY HTN-3 Investigators. A controlled trial of renal denervation for resistant hypertension. N Engl J Med. 2014 Apr 10;370(15):1393-401. doi: 10.1056/NEJMoa1402670. Epub 2014 Mar 29. PMID 24678939
- [Background] D'Elia E, Pascale A, Marchesi N, Ferrero P, Senni M, Govoni S, Gronda E, Vanoli E. Novel approaches to the post-myocardial infarction/heart failure neural remodeling. Heart Fail Rev. 2014 Sep;19(5):611-9. doi: 10.1007/s10741-013-9415-6. PMID 24292688